CLINICAL TRIAL: NCT00206258
Title: The Role of Amylin and Glucagon in the Management of Normalizing Glucose Excursions in Children With Type 1 Diabetes
Brief Title: The Role of Amylin and Glucagon in T1DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sponsored Programs, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-11741
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; hypoglycemia; hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia | interventions — pramlintide; Glucagon

INTERVENTIONS:
Drug: Pramlintide and glucagon

SUMMARY:
The purpose of this study is to see if giving pramlintide and insulin before a meal would lower high blood sugar and if a glucagon (a naturally made hormone in the body but reduced in diabetes and its role is in prevention of low blood sugar) shot given in the late "after meal" time would prevent low blood sugar. The studies outlined in this proposal might help in developing new treatment options to target "after meal" high blood sugar and before meal low blood sugar in children. This would possibly help improve overall blood sugar control and prevent the long-term complications of diabetes.

DETAILED DESCRIPTION:
Objective: To develop a new treatment approach in the prevention of hypo and hyperglycemia in children with type 1diabetes.

Background/Rationale: The diabetes control and complications trial (DCCT) showed that improving blood sugar control for individuals with type 1 diabetes (T1DM) stopped or delayed the onset of long-term complications. As a result of the study, intensive management to control blood sugar and glycosylated hemoglobin as near to normal as safely as possible is advocated. However, hypoglycemia was increased 3 fold in the DCCT study and is the major limiting factor in gaining "tight" control of blood sugar in T1DM.

Description of Project: In health individuals, "after meal" blood sugar level is very carefully controlled. Insulin (the hormone that lowers blood sugar) and glucagon (the hormone that raises blood sugar) play a key role in maintaining this careful balance. Recently we understand that a hormone called amylin also contributes to this careful after meal blood glucose balance. Amylin in the immediate after meal period works by reducing glucagon, which in turn reduces the liver releasing stored sugar into the blood stream.

In T1DM, there is the lack of insulin and failure of glucagon suppression leading to hyperglycemia immediately following when food is eaten. Also, glucagon is not regulated correctly after a meal. The glucagon normally produced by the body does not increase in response to hypoglycemia thus interfering with the delicate balance between glucose production and glucose used. Therefore, it is difficult to get normal blood sugar when someone has type1 diabetes.

Currently, the treatment for mild to moderate hypoglycemia causing a sudden feeling of racing heart, feeling sweaty, weak or hungry is to eat or drink carbohydrate in the awake person. Severe hypoglycemia (unconsciousness due to low blood sugar) is treated with a glucagon shot. Unfortunately, there are no treatments to prevent mild or severe hypoglycemia.

The purpose of this study is to see if giving pramlintide (manmade amylin) and insulin before a meal would lower hyperglycemia and if a glucagon shot given in the late "after meal" time would prevent hypoglycemia and allow the blood sugar levels to improve in people with T1DM. The studies outlined in this proposal might help in developing new treatment options to target "after meal" hyperglycemia high blood glucose and before meal hypoglycemia in children. This study for the first time will investigate the role of glucagon in the causation of hyperglycemia and its role in the prevention of hypoglycemia.

Relevance to Type 1 diabetes: Using naturally occurring hormones that are dysregulated or deficient in T1DM we wish to restore normal glucose concentration in T1DM. Such treatment if successful would be a major breakthrough in the prevention of hyper and hypoglycemia and in decreasing both short and long-term complications associated with T1DM.

ELIGIBILITY:
Inclusion Criteria:

1. Age >12 years < 19 years
2. Have diabetes for at least 2 years and in good control (HbA1C < 8%).
3. Be on continuous subcutaneous insulin infusion using an insulin pump.
4. Subjects must be otherwise healthy except for their T1DM and treated for hypothyroidism.
5. Menstruating women must have negative pregnancy test.
6. Hemoglobin equal to or > than 12 g/dL before each study.
7. Weight more than 44 kg.

Exclusion Criteria:

1. Age >18 or < 12 y at the time of study
2. Any chronic disease (leukemia, asthma, inflammatory bowel disease, cystic fibrosis, juvenile rheumatoid arthritis, etc that directly, or as a result of treatment, directly or indirectly affect glucose homeostasis
3. Hemoglobin less than 12 g/dl (If before any of the studies the hemoglobin is lower than 12 g/dl, subjects will be excluded from further studies)
4. Lack of a supportive family environment
5. Positive pregnancy test in menstruating young women
6. Evidence or history of chemical abuse
7. Hgb A1c >8.0 % in a diabetic subject
8. BMI > 90 % tile for age or < 10 % tile for age
9. Allergy to local anesthetics (ELAMAX Cream)
10. Weight less than 44 kg
11. Children of staff members

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2002-07; Study Completion 2005-08

PRIMARY OUTCOMES:
Area under the curve for glucose

SECONDARY OUTCOMES:
Glucagon and gastric emptying

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Heptulla, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Result] Heptulla RA, Rodriguez LM, Bomgaars L, Haymond MW. The role of amylin and glucagon in the dampening of glycemic excursions in children with type 1 diabetes. Diabetes. 2005 Apr;54(4):1100-7. doi: 10.2337/diabetes.54.4.1100. PMID 15793249
- See also: Learn about the physiology of amylin — http://amylin.org